CLINICAL TRIAL: NCT00524654
Title: The Effects of Cervical Spine Manipulation On Postural Control
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: SR0411060017
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Posture
Keywords: To determine the effects of cervical spine manipulation on postural control.

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Procedure: HVLA chiropractic manipulation

SUMMARY:
The purpose of this study is to test the effect of high velocity low amplitude (HVLA) chiropractic cervical manipulation on the patient's postural control as measured by a force plate.

ELIGIBILITY:
Inclusion Criteria:

* Students
* Normal healthy adults

Exclusion Criteria:

* Previous or ongoing foot, ankle, or hip problems
* Experiencing vertigo, visual difficulties and other disorders that would make it difficult to balance for a set period of time.
* Anyone with high risk for injury due to cervical manipulation
* Anyone with training in areas of activity that require superior balance
* Body mass index over 30

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodger Tepe, PhD, Principal Investigator — Logan College
Locations (1):
- Logan College, Chesterfield, Missouri, United States